CLINICAL TRIAL: NCT02952950
Title: Is it Possible to Prolong the Duration of Exclusive Breastfeeding in Premature Infants? a Prospectivt Study
Brief Title: Is it Possible to Prolong the Duration of Breastfeeding in Premature Infants? a Prospectivt Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Diana Skaaning, Principal Investigator, Hvidovre University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: H-16000621
Record Dates: First submitted 2016-11-01; First posted 2016-11-02 (Estimated); Last update posted 2019-09-25 (Actual); Status verified 2018-02

CONDITIONS: Breast Feeding; Premature Birth
Keywords: Intra Oral Vacuum; protein content breastmilk
MeSH Terms: conditions — Breast Feeding; Premature Birth

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oralstimulation (Other): Infants whose mothers is included in the cohort is randomized to receive oral stimulation when the infant's postnatal age is at least 32 + 0 weeks, as it is the time when the infant is able to coordinate sucking and swallowing reflex
  Interventions: Other: Oralstimulation
- Controlgroup (No Intervention): Families in the control group is not seeing the oralstimulation movie, do not receive the script or the supervision of occupational therapists and these infants do not get oral stimulation. Both groups receive instructions after usual practice i.e. guidance and elements that promote breastfeeding example, skin to skin contact and compression.

INTERVENTIONS:
Other: Oralstimulation — The intervention group granted in total 1 hour instructions in a program of oral stimulation by one of two occupational therapists with experience in oral stimulation of preterm infants. The first guidance for parents has duration of approximately half an hour and then follow-up once or twice, depending on the needs of the family. To maintain consistent intervention over time is the program of oral stimulation written in a script, where the family also must record the following variables: date and time of oral stimulation. In occupational therapy the guidance and in the script examines the signs that the infant exhibits when it is ready / not ready for stimulation. The family also sees a movie where these signs and the program of oral stimulation review auditory and visual.
  Arms: Oralstimulation

SUMMARY:
In this project three studies examined two possible explanations and one possible preventive intervention to early cessation of exclusively breastfeeding in premature infants.

Study 1 The content of protein in the milk of mothers, who delivers prematurely, is about a third higher than in the milk from the mother who delivers on time. The nutritional composition changes over time and the content of protein decrease. Therefore the premature infant is at risk of protein deficiency. While the infant is feeding by tube this decreasing content of protein can made up by adding, while it is more difficult when the infant is exclusively breastfeeding. The hypothesis is that reduced protein content in breast milk is associated to a fewer number of days where the premature infant is exclusively breastfed.

Study 2 The premature infant is characterized with immature muscle with a low tension and therefore, a low ability to eat its needs by breastfeeding the first period. The transfer of milk from mother to child is an interaction between the mothers and her milk ejection reflex that establish a positive pressure on the milk and the child that have to establish a vacuum. The hypothesis is that the premature infants suction power is too weak to establish sufficient intraoral vacuum to ensure milk transfer from the breast to the infant and it can be related to a fewer number of days where the infant is exclusively breastfed.

Study 3 The premature infants low muscle tone and its immaturity also influence on the organization and the quality of movements, marked as neuro motor processes. These processes form the oral motor base supporting movement which involves the infant ability to establish vacuum. The hypothesis is that Oral Stimulation for a specific program in 5 minutes before the minimum 2 meals per. day for at least 14 days increases the preterm infant's ability to create intra oral vacuum and thus the power to transfer milk from the breast, thereby extending the number of days when the infant is exclusively breastfed.

200 infants are included consecutively, as a recurring cohort in all 3 studies. In Study 1 the mothers' milk is analyzed in order to the content of protein. In Study 2 the infant suction is assessed by vacuum measurement. In study 3 the families are randomized to an intervention or control group and parents off 100 infants are guided by occupational therapists in a program of oral stimulation of their child.

DETAILED DESCRIPTION:
The purpose of this project, which consists of three studies, is to investigate whether insufficient protein in breastmilk and / or inadequate intra oral vacuum of the infant can explain early breastfeeding cessation in the premature infant. Furthermore to test whether the breastfeeding period may be extended by oral stimulation.

The rate of breastfeeding in mothers of infants born prematurely is lower than in mothers who give birth on time. A Danish survey shows that about 70% of premature are on exclusive breastfeeding at discharge and that this rate is decreasing to about 30% six weeks after discharge. Breastmilk is the healthiest nutrition for the newborn and based on WHO's strategy for the feeding of infants Board of Health recommends that newborn infants, including premature, as far as possible are exclusively breastfed for six months. Exclusively breastfeeding means that the infant only gets the breastmilk of the mother. Exclusively breastfeeding has health implications for both mother and infant. Breastfeeding reduces lactation incidence of infectious diseases, improves cognitive development and visual function in the infant and reduces the risk of developing later obesity. In addition, the level of immune protective factors and anti-inflammatory elements is high in the mother's milk to the preterm infant and therefore reduce the infant's increased risk of early and severe infections, and death late effects. Furthermore, breastfeeding may reduce the risk of premature infant's abnormal vessel growth in the eye, and appears to have a protective effect on the disease being of significant excess mortality primarily attack the intestines of the preterm infant (necrotizing enterocolitis).

Problem Area / factors in milk composition with the importance of breastfeeding Breastmilk contains the necessary nutritional components and energy that the infant needs. Therefore, the milk of the mother delivering early have a higher content of fat and protein, and thereby a higher level of energy comparing with the milk from the mother who have given birth to term. The content of protein in the milk of the mother who gives birth prematurely is about 12 grams per liter and thus approximately one-third higher than that from the mother who gives birth on time. The nutritional composition of breastmilk vary considerably over time and the content of protein is decreasing why the premature infant are at risk of protein deficiency and thereby insufficient growth. During the hospital stay, and while the infant are feed by tube this decreasing protein content are made up by adding, while it is more difficult when the infant breastfeed exclusively. Protein is important for the infant's growth and strength and a local statement from Hvidovre Hospital found that 18% of all hospitalized preterm infants in 2014 were added additional protein to breastmilk, because growth was not sufficient. The question is whether reduced protein content in breastmilk has a correlation with the number of days where preterm infants are exclusively breastfed?

Problem Area / intra oral vacuum strength of the infant with significance for breastfeeding The period from birth to the premature infant feed exclusively at the breast without supplementary tube feeding varies from weeks to months, depending on how early the infant is born. The premature infant is characterized as being immature and with low muscle tone and therefore, a decreased ability to breastfeed the first time. The transfer of milk from mother to infant is an interaction between the mother and her milk ejection reflex creates a positive pressure on the milk and the infant creates a vacuum. If the infant not create a vacuum at the back of the mouth, the nipple of the mother is just pushed together and the infant is not transferred milk from the breast to the oral cavity. The amount of milk is regulated in relation to demand and a weak or shortage of vacuum will cause a shortage of milk transfer, which in turn physiologically will lead to less milk production and thereby decreasing amount. Studies that investigates this process and measured intra oral vacuum, shows all the importance of the infant's contribution by milk transfer, but does not answer to the extent the premature infants ability to create vacuum importance of breastfeeding establishment and maintaining. The question is whether the premature infants sucking strength is too weak to establish sufficient intraoral vacuum to ensure milk transfer from the breast to the infant and it can be related to a fewer number of days where the infant is exclusively breastfed.

In addition to the premature infants muscle tone has its immaturity also affect the organization and quality of body movements. Organization and quality in the movements may be referred to neuro motor processes and form among others the oral motor base supporting the movements involving the infant's ability to create vacuum. The processes preceding the creation of vacuum and studies have shown that by early intervention with oral stimulation in the form of stimulation of the nerves and muscles in and around the mouth, it can be oral motor basis strengthened. Studies where the infant carefully is stimulated with a finger, showing that the premature infant's muscles and sucking reflex can be influenced so that it is able to suck a larger volume in a shorter time in the bottle compared to the infant that is not stimulated orally. This presents an opportunity to influence the premature infant´s strength and maybe increase the ability to create intra oral vacuum affected by oral stimulation as a skill the infant preserves. The question is whether oral stimulation can increase the premature infant's ability to create vacuum and thus increase the power to transfer milk from the breast and thereby extending the number of days when with exclusively breastfed? The 3 studies are based on the same cohort. The cohort is identified and recruited at the Neonatal Intensive Care Unit at Hvidovre Hospital and relevant families where the mother delivers prematurely are included consecutively in accordance to the inclusion and exclusion criteria. The cohort will be demographically representative of everyday life in clinical practice with various family formation, education levels and socio-economic background conditions.

Power calculations are based primary outcome: exclusively breastfeeding duration and made to show effect on exclusively breastfeeding duration between the intervention- and the control group. Requirements for power calculation are a mean value of the vacuum set at 100% with a standard deviation (SD) of 26%. To detect the smallest clinically relevant difference of 13%, equivalent to half a SD and with an expected drop out of 20%, which included 200 infants (100 infants in each group) in the study (alpha = 0.05 and beta = 0.1 ). There hospitalized annually on average 300 preterm infants in the neonatal section. It is expected about 100 infants to meet the criteria for inclusion, thus achieved at approximately 2 year.

By inclusion the family is anonymized by allocating an ID number. When multiple assigned each infant this ID number and a one of letters a, b or c. All data and all measurements is obtained / made and recorded as far as possible of the project manager or alternatively the project nurse.

6 weeks after the date for the expected terminator date either the family are visiting the Neonatal section or the project manager/project nurse visiting the family in order to a status of breastfeeding, vacuum measurement and the infant's growth. In addition the family is contact by telephone the week in which the infant's postnatal age is 6 months. Here is recorded breastfeeding status, the time of any termination of exclusive breastfeeding and the infant's weight at GP visit 5 month old. The infant's growth is defined by its naked weight, Length and head circumference. Previous studies show a number of factors which affect breastfeeding duration. Features concerning socio-demographic background variables, perinatal and psychosocial conditions will gathered by the project manager or project nurse using a questionnaire in an interview with the family and form data in the analyzes. Participation in the project is safe and not associated with risk or discomfort for either mother or infant.

STUDY 1 / PROTEIN IN BREASTMILK Data are obtained in the human milk section at the hospital. Volume is obtained in milliliter (ml.) and protein content in gram pr. 100 ml. by using Miris Human Milk Analyzer according to the usual practice. Miri is the only European equipment that analyzes human milk. The test sample is 10 milliliters and the result given within a minute and logged into the machine and then transferred to the project database. When the mother is exclusively breastfeeding, we ask for 10 ml. Manual hand compressed breast milk. The analyzed milk can´t be reused and is therefore destroyed.

STUDY 2 / WEEK STRENGTH ASSESSMENT BY VACUUM MEASUREMENT Sucking strength of the premature infant is defined as the ability to create intra oral vacuum during sucking.

The intra oral vacuum of the premature infant is assessed by measuring the vacuum in the unit of mBar and are primary made by the project manager which is blinded to know if the infant has received oral stimulation or not. The measurement is made when the infant is awake and show readiness to suck. For vacuum measurement is a manometer selected with a bottle pacifier, which fits a Calmaflaske made by the firm Medela. The pacifier is shaped and is similar in function a breast and extra small so that it matches the premature mouth of a premature infant. As in a completely closed system the sucking of the infant is registered on this connected manometer. In order to obtain a measure of reproducibility of the method all vacuum measurements is carried out at 3 consecutive measurements. The advantage of the 3 measurements within a short time is to determine the intra-individual variability, but only if the infant is motivated and show redlines for measurement 3 times. The equipment is developed in cooperation with the Technical University of Denmark.

STUDY 3 / randomized INTERVENTION STUDY / ORAL STIMULATION Infants whose mothers is included in the cohort is randomized to receive / not receive oral stimulation when the infant's postnatal age is at least 32 + 0 weeks, as it is the time when the infant is able to coordinate sucking and swallowing reflex. In multiple birth all infants is randomized to the same group. The list is generated block randomized in blocks of 10

Families were randomized to the intervention group granted in total one hour instructions in a program of oral stimulation by one of two occupational therapists with experience in oral stimulation of preterm infants. The program is in collaboration with the project team developed and described by the Department of Physiology and Occupational therapy at Hvidovre Hospital. The first guidance for parents has duration of approximately half an hour and then follow-up once or twice, depending on the needs of the family. To maintain consistent intervention over time is the program of oral stimulation written in a script, where the family also must record the following variables: date and time of oral stimulation. In occupational therapy the guidance and in the script examines the signs that the infant exhibits when it is ready / not ready for stimulation. The family also sees a movie where these signs and the program of oral stimulation review auditory and visual. Families in the control group is not seeing the movie, do not receive the script or the supervision of occupational therapists and these infants do not get oral stimulation. Both groups receive instructions after usual practice i.e. guidance and elements that promote breastfeeding example, skin to skin contact and compression.

ELIGIBILITY:
Inclusion Criteria:

* mothers: with premature infant i.e. the infant's gestational age is equal to or maximum of 36 + 6
* intend to breastfeed.
* The mother or father / other primary caregiver understand Danish, Norwegian, Swedish or English.

Exclusion Criteria:

* mothers: will not / can´t breastfeed because of illness or abuse such as: HIV and drugs.
* In addition, if the infant has a disability which makes it difficult to breastfeeding or if the infant is physiologically unstable, for example due to reduced lung function.

Max Age: 37 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 211 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
Duration of Breastfeeding | 6 month
  Exclusively breastfeeding duration measured in number of whole days and defined as the infant is exclusively fed with breastmilk

SECONDARY OUTCOMES:
Content of protein in breastmilk | 6 weeks after the terminator date
  Protein content are examined once a week as long the family is hospitalized and 6 weeks after the terminator date.
Intra Oral Vacuum | 6 weeks after the terminator date
  Intra oral vacuum are examined once a week as long the family is hospitalized and 6 weeks after the terminator date.

CONTACTS AND LOCATIONS:
Overall Officials: Ole Pryds, Dr.MedShi, Study Chair — Regionshospitalet Randers Paediatric Department
Locations (1):
- Paediatric Department section Neonatology, Hvidovre, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Maastrup R, Hansen BM, Kronborg H, Bojesen SN, Hallum K, Frandsen A, Kyhnaeb A, Svarer I, Hallstrom I. Factors associated with exclusive breastfeeding of preterm infants. Results from a prospective national cohort study. PLoS One. 2014 Feb 19;9(2):e89077. doi: 10.1371/journal.pone.0089077. eCollection 2014. PMID 24586513
- [Background] Pimenta HP, Moreira ME, Rocha AD, Gomes SC Jr, Pinto LW, Lucena SL. Effects of non-nutritive sucking and oral stimulation on breastfeeding rates for preterm, low birth weight infants: a randomized clinical trial. J Pediatr (Rio J). 2008 Sep-Oct;84(5):423-7. doi: 10.2223/JPED.1839. English, Portuguese. PMID 18923786
- [Background] Wambach K, Riordan J, redaktører. Breastfeeding and human lactation. Fifth edition. Burlington, Massachusetts: Jones & Bartlett Learning; 2015.
- [Background] Cope MB, Allison DB. Critical review of the World Health Organization's (WHO) 2007 report on 'evidence of the long-term effects of breastfeeding: systematic reviews and meta-analysis' with respect to obesity. Obes Rev. 2008 Nov;9(6):594-605. doi: 10.1111/j.1467-789X.2008.00504.x. Epub 2008 Jun 12. PMID 18554244
- [Background] Vohr BR, Poindexter BB, Dusick AM, McKinley LT, Higgins RD, Langer JC, Poole WK; National Institute of Child Health and Human Development National Research Network. Persistent beneficial effects of breast milk ingested in the neonatal intensive care unit on outcomes of extremely low birth weight infants at 30 months of age. Pediatrics. 2007 Oct;120(4):e953-9. doi: 10.1542/peds.2006-3227. PMID 17908750
- [Background] Cristofalo EA, Schanler RJ, Blanco CL, Sullivan S, Trawoeger R, Kiechl-Kohlendorfer U, Dudell G, Rechtman DJ, Lee ML, Lucas A, Abrams S. Randomized trial of exclusive human milk versus preterm formula diets in extremely premature infants. J Pediatr. 2013 Dec;163(6):1592-1595.e1. doi: 10.1016/j.jpeds.2013.07.011. Epub 2013 Aug 20. PMID 23968744
- [Background] Groh-Wargo S, Sapsford A. Enteral nutrition support of the preterm infant in the neonatal intensive care unit. Nutr Clin Pract. 2009 Jun-Jul;24(3):363-76. doi: 10.1177/0884533609335310. PMID 19483066
- [Background] Smith JP, Harvey PJ. Chronic disease and infant nutrition: is it significant to public health? Public Health Nutr. 2011 Feb;14(2):279-89. doi: 10.1017/S1368980010001953. Epub 2010 Jul 13. PMID 20624333
- [Background] Hylander MA, Strobino DM, Pezzullo JC, Dhanireddy R. Association of human milk feedings with a reduction in retinopathy of prematurity among very low birthweight infants. J Perinatol. 2001 Sep;21(6):356-62. doi: 10.1038/sj.jp.7210548. PMID 11593368
- [Background] McGuire W, Anthony MY. Donor human milk versus formula for preventing necrotising enterocolitis in preterm infants: systematic review. Arch Dis Child Fetal Neonatal Ed. 2003 Jan;88(1):F11-4. doi: 10.1136/fn.88.1.f11. PMID 12496220
- [Background] Agostoni C, Buonocore G, Carnielli VP, De Curtis M, Darmaun D, Decsi T, Domellof M, Embleton ND, Fusch C, Genzel-Boroviczeny O, Goulet O, Kalhan SC, Kolacek S, Koletzko B, Lapillonne A, Mihatsch W, Moreno L, Neu J, Poindexter B, Puntis J, Putet G, Rigo J, Riskin A, Salle B, Sauer P, Shamir R, Szajewska H, Thureen P, Turck D, van Goudoever JB, Ziegler EE; ESPGHAN Committee on Nutrition. Enteral nutrient supply for preterm infants: commentary from the European Society of Paediatric Gastroenterology, Hepatology and Nutrition Committee on Nutrition. J Pediatr Gastroenterol Nutr. 2010 Jan;50(1):85-91. doi: 10.1097/MPG.0b013e3181adaee0. PMID 19881390
- [Background] Sakalidis VS, McClellan HL, Hepworth AR, Kent JC, Lai CT, Hartmann PE, Geddes DT. Oxygen Saturation and Suck-Swallow-Breathe Coordination of Term Infants during Breastfeeding and Feeding from a Teat Releasing Milk Only with Vacuum. Int J Pediatr. 2012;2012:130769. doi: 10.1155/2012/130769. Epub 2012 May 9. PMID 22844300
- [Background] Boiron M, Da Nobrega L, Roux S, Saliba E. Pharyngeal swallowing rhythm in response to oral sensorimotor programs in preterm infants. J Neonatal Nurs. 2009;15(4):123-8.
- [Background] Geddes DT, Sakalidis VS, Hepworth AR, McClellan HL, Kent JC, Lai CT, Hartmann PE. Tongue movement and intra-oral vacuum of term infants during breastfeeding and feeding from an experimental teat that released milk under vacuum only. Early Hum Dev. 2012 Jun;88(6):443-9. doi: 10.1016/j.earlhumdev.2011.10.012. Epub 2011 Nov 26. PMID 22119233
- [Background] Morris SE. Development of oral-motor skills in the neurologically impaired child receiving non-oral feedings. Dysphagia. 1989;3(3):135-54. doi: 10.1007/BF02407132. PMID 2517923
- [Background] Harding C. An evaluation of the benefits of non-nutritive sucking for premature infants as described in the literature. Arch Dis Child. 2009 Aug;94(8):636-40. doi: 10.1136/adc.2008.144204. PMID 19628881
- [Background] Lessen BS. Effect of the premature infant oral motor intervention on feeding progression and length of stay in preterm infants. Adv Neonatal Care. 2011 Apr;11(2):129-39. doi: 10.1097/ANC.0b013e3182115a2a. PMID 21730902
- [Background] Neiva FC, Leone CR. [Sucking in preterm newborns and the sucking stimulation]. Pro Fono. 2006 May-Aug;18(2):141-50. doi: 10.1590/s0104-56872006000200003. Portuguese. PMID 16927619
- [Background] Ratnovsky A, Carmeli YN, Elad D, Zaretsky U, Dollberg S, Mandel D. Analysis of facial and inspiratory muscles performance during breastfeeding. Technol Health Care. 2013;21(5):511-20. doi: 10.3233/THC-130749. PMID 24177309
- [Background] Boiron M, Da Nobrega L, Roux S, Henrot A, Saliba E. Effects of oral stimulation and oral support on non-nutritive sucking and feeding performance in preterm infants. Dev Med Child Neurol. 2007 Jun;49(6):439-44. doi: 10.1111/j.1469-8749.2007.00439.x. PMID 17518930
- [Background] Fucile S, Gisel EG, McFarland DH, Lau C. Oral and non-oral sensorimotor interventions enhance oral feeding performance in preterm infants. Dev Med Child Neurol. 2011 Sep;53(9):829-835. doi: 10.1111/j.1469-8749.2011.04023.x. Epub 2011 Jun 27. PMID 21707601
- [Background] Fucile S, Gisel EG, Lau C. Effect of an oral stimulation program on sucking skill maturation of preterm infants. Dev Med Child Neurol. 2005 Mar;47(3):158-62. doi: 10.1017/s0012162205000290. PMID 15739719
- [Background] Fucile S, McFarland DH, Gisel EG, Lau C. Oral and nonoral sensorimotor interventions facilitate suck-swallow-respiration functions and their coordination in preterm infants. Early Hum Dev. 2012 Jun;88(6):345-50. doi: 10.1016/j.earlhumdev.2011.09.007. Epub 2011 Sep 29. PMID 21962771
- [Background] Maastrup R, Hansen BM, Kronborg H, Bojesen SN, Hallum K, Frandsen A, Kyhnaeb A, Svarer I, Hallstrom I. Breastfeeding progression in preterm infants is influenced by factors in infants, mothers and clinical practice: the results of a national cohort study with high breastfeeding initiation rates. PLoS One. 2014 Sep 24;9(9):e108208. doi: 10.1371/journal.pone.0108208. eCollection 2014. PMID 25251690
- [Background] Flacking R, Ewald U, Starrin B. "I wanted to do a good job": experiences of 'becoming a mother' and breastfeeding in mothers of very preterm infants after discharge from a neonatal unit. Soc Sci Med. 2007 Jun;64(12):2405-16. doi: 10.1016/j.socscimed.2007.03.008. Epub 2007 Apr 10. PMID 17428597
- [Background] Aizawa M, Mizuno K, Tamura M. Neonatal sucking behavior: comparison of perioral movement during breast-feeding and bottle feeding. Pediatr Int. 2010 Feb;52(1):104-8. doi: 10.1111/j.1442-200X.2009.02914.x. Epub 2009 Jun 22. PMID 19552641
- [Background] Geddes DT, Kent JC, Mitoulas LR, Hartmann PE. Tongue movement and intra-oral vacuum in breastfeeding infants. Early Hum Dev. 2008 Jul;84(7):471-7. doi: 10.1016/j.earlhumdev.2007.12.008. Epub 2008 Feb 11. PMID 18262736